CLINICAL TRIAL: NCT02454270
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of Duvortuxizumab, A Humanized CD19 x CD3 Dual-Affinity Re-Targeting (DART®) Protein in Subjects With Relapsed or Refractory B-cell Malignancies
Brief Title: A Dose Escalation Study of Duvortuxizumab in Participants With Relapsed or Refractory B-cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recent advances in the treatment of B cell malignancies resulting in new treatments being approved for marketing and many others in late stage development
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107241; 2015-000485-63 (EudraCT Number); 64052781LYM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-05-06; First posted 2015-05-27 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: First-in-Human; B-Cell Chronic Lymphocytic Leukemia; Diffuse Large-Cell Lymphoma; Follicular Lymphoma; Mantle-Cell Lymphoma; Acute Lymphoid Leukemia; Dose Escalation Study; Duvortuxizumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Dose Escalation: Participants With Certain B-Cell Malignancies (Experimental): During accelerated dose titration in Group 1, participant will receive duvortuxizumab starting at 0.5 nanogram per kilogram (ng/kg) for biweekly dosing. Dose will be increased by half logarithmic steps in subsequent Dose Level (DL). After safety stopping criteria are met, Dose Escalation (DE) in Group 1 will transition to 3+3 design, and will continue until the Maximum tolerated Dose (MTD) is defined. DE in Groups 2 and 3 will follow 3+3 design, begin after initial dose level in Group 1 is deemed safe and recommended phase 2 doses (RP2D) for Part 1 of study can be decided. Duvortuxizumab at a starting dose of 50 ng/kg weekly will also be investigated in Group 1 and will follow 3+3 study design continue until the MTD or Maximum administered dose (MAD) is reached. Disease-specific dose escalation in Group 2 and 3 will not be initiated until dose in Group 1 is determined safe.
  Interventions: Drug: Part 1 (Dose Escalation): Duvortuxizumab
- Dose Expansion: Diffuse-Large B-Cell Lymphoma Participants (Experimental): Participants with Diffuse-Large B-Cell Lymphoma (DLBCL) will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) either with or without a priming dose.
  Interventions: Drug: Part 2 (Dose Expansion): Duvortuxizumab
- Dose Expansion: Follicular Cell Lymphoma Participants (Experimental): Participants with Follicular Cell Lymphoma (FL) will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) either with or without a priming dose.
  Interventions: Drug: Part 2 (Dose Expansion): Duvortuxizumab
- Dose Expansion: Mantle Cell Lymphoma Participants (Experimental): Participants with Mantle Cell Lymphoma (MCL) will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) either with or without a priming dose.
  Interventions: Drug: Part 2 (Dose Expansion): Duvortuxizumab
- Dose Expansion: Chronic Lymphocytic Leukemia Participants (Experimental): Participants with Chronic Lymphocytic Leukemia (CLL) will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) either with or without a priming dose.
  Interventions: Drug: Part 2 (Dose Expansion): Duvortuxizumab
- Dose Expansion: Acute Lymphoblastic Leukemia Participants (Experimental): Participants with Acute Lymphoblastic Leukemia (ALL) will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) either with or without a priming dose.
  Interventions: Drug: Part 2 (Dose Expansion): Duvortuxizumab

INTERVENTIONS:
Drug: Part 1 (Dose Escalation): Duvortuxizumab — Participants currently enrolled in the study will continue to receive duvortuxizumab every 14 days (biweekly dosing) in each 28 -day cycle as an intravenous infusion. In the priming dose regimen, a priming dose will be administered on Day 1 followed by full doses on Day 8 and Day 22, of a 35-day Cycle 1, and then every 14 days in each subsequent 28-day cycle. The cohorts will be opened where participants will receive duvortuxizumab every 7 days (for investigating weekly dosing schedule) in each 28-day cycle as an intravenous infusion. In the priming dose regimen, a priming dose will be administered on Day 1 followed by full doses on Day 8, Day 15, Day 22, and Day 28 of a 35-day Cycle 1, and then every 7 days in each subsequent 28-day cycle.
  Arms: Dose Escalation: Participants With Certain B-Cell Malignancies
Drug: Part 2 (Dose Expansion): Duvortuxizumab — Participants will receive intravenous infusion of duvortuxizumab at the recommended Phase 2 dose (RP2D) defined in Part 1 for their disease type either with or without a priming dose.
  Arms: Dose Expansion: Acute Lymphoblastic Leukemia Participants; Dose Expansion: Chronic Lymphocytic Leukemia Participants; Dose Expansion: Diffuse-Large B-Cell Lymphoma Participants; Dose Expansion: Follicular Cell Lymphoma Participants; Dose Expansion: Mantle Cell Lymphoma Participants

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dose-limiting toxicities (any harmful effect of a drug) (DLT), maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D) and preliminary clinical activity of duvortuxizumab when administered intravenously to participants with relapsed or refractory B-cell malignancies [diffuse-large B cell lymphoma (DLBCL), follicular lymphoma (FL), mantle-cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), and acute lymphoblastic leukemia (ALL)].

DETAILED DESCRIPTION:
This first in human study consists of 2 parts: a) The dose escalation part and b) The dose expansion part. This is an openlabel (all participants know the identity of the intervention), multicenter (more than one study site) study to evaluate the safety, establish a recommended Phase 2 dose (RP2D), and to determine the preliminary efficacy of duvortuxizumab in participants with relapsed or refractory B cell malignancies. The dose escalation part of the trial (Part 1) will be comprised of 3 different patient groups based on disease indication: Group 1 (DLBCL, FL, MCL); Group 2 (CLL); Group 3 (ALL). The duvortuxizumab dosing will be done on biweekly and weekly basis. Duvortuxizumab weekly escalating dosing will be investigated. Dose escalation will begin with Group 1 and will initially follow an accelerated dose titration design, followed by a traditional 3+3 design. At each dose escalation level the treatment of the second participant should be initiated after at least 72 hours of observation after the start of the first duvortuxizumab dose of the first participant. Dose escalation in Groups 2 and 3 will follow a 3+3 design and will begin after the initial dose level in Group 1 is deemed safe. Participants [Group 1 (DLBCL, FL, MCL), Group 2 (CLL) Group 3 (ALL)] are enrolled into cohorts of increasing dose levels of duvortuxizumab administered in 28 day treatment cycles. Up to 3 RP2Ds may be determined in Part 1 (one RP2D for Group 1, one RP2D for Group 2, and one RP2D for Group 3). In the cohort expansion part of the trial (Part 2), participants with relapsed or refractory B cell malignancies (DLBCL, FL, MCL, CLL and ALL) will be enrolled according to tumor type in up to 5 cohorts and receive duvortuxizumab at the RP2D determined in Part 1 for their disease type. The study consists of 3 periods: Screening period (up to 28 days prior to the first dose of study drug); Treatment period [first dose of study drug until the End of Treatment Visit (within 30 days after the last dose)]; and follow up period [End of Treatment Visit and continue until death, lost to follow up, consent withdrawal, or study end (as determined by the sponsor), whichever occurs first]. Number of participants who achieve an overall response in each Dose Expansion cohort will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Participants must meet protocol specified hematology and chemistry lab parameters criteria
* Histological confirmation of disease with documented disease relapse after the last therapy requiring treatment per the treating physician. Participants with lymphoma must have at least 1 measurable site of disease (Part 2 only). In addition, B-cell malignancy disease-specific criteria specified in the protocol must also be met
* A woman of childbearing potential must have a negative highly sensitive serum [beta-human chorionic gonadotropin (β-hCG)] or urine pregnancy test at (minimum sensitivity 25 International units (IU)/ liter (L) or equivalent units of HCG) within 7 days prior to the first dose of study drug
* A woman must agree to use an effective method of birth control and agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after receiving the last dose of study drug
* A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (eg, condom with spermicidal foam/gel/film/cream/suppository), man who is sexually active with a woman who is pregnant must use a condom and men must agree not to donate sperm for 90 days after the last dose of study drug
* Each participant (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Consent is to be obtained prior to the initiation of any study related tests or procedures that are not part of standard of care for the participant's disease

Exclusion Criteria:

* History of, or known central nervous system (CNS) involvement caused by the underlying B-cell malignancy or prior history of National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) Grade greater than or equal to >= 3 drug-related CNS toxicity. Participants with signs or symptoms of CNS involvement should have a computed tomography (CT) or magnetic resonance imaging (MRI)
* History of or known or suspected autoimmune disease (exception: vitiligo, resolved childhood atopic dermatitis, and history of Grave's disease that is euthyroid clinically and by laboratory testing at Screening)
* Prior allogeneic hematopoietic stem-cell transplant for participants with DLBCL, FL, MCL, and CLL only. Prior allogenic hematopoietic stem-cell transplant is permitted for participants with ALL
* Prior solid organ transplantation
* Prior treatment with a therapeutic agent targeting CD19 and/or CD3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Part 1: Recommended Phase 2 Dose (RP2D) of Duvortuxizumab | Approximately 15 months
  The RP2D will be determined based on safety, clinical activity, pharmacokinetics, and pharmacodynamics in participants with relapsed or refractory B cell malignancies [diffuse large B cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL) and acute lymphoblastic leukemia (ALL)].
Part 2: Number of Participants With Overall Response Rate (ORR) | Approximately 2 Years
  The ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR) per criteria for response assessment of Non Hodgkin Lymphomas (NHL) or International Workshop on Chronic Lymphocytic Leukemia (IWCLL), or complete response (CR), complete response with partial hematologic recovery (CRp), or complete response with incomplete recovery of counts (CRi) per response criteria for acute lymphoblastic leukemia (ALL).

SECONDARY OUTCOMES:
Part 1 and 2: Area Under the Curve From Time Zero to End of Dosing Interval (AUC tau) of Duvortuxizumab | Approximately 2 Years
  The AUC tau is the area under the serum concentration versus time curve during a dose interval time period (tau).
Part 1 and 2: Maximum Serum Concentration (Cmax) of Duvortuxizumab | Approximately 2 Years
  The Cmax is the maximum observed serum concentration of duvortuxizumab.
Part 1 and 2: Half-Life (t1/2) of Duvortuxizumab | Approximately 2 Years
  The t(1/2) is defined as 0.693/Lambda (z)
Part 1 and 2: Total Systemic Clearance (CL) of Duvortuxizumab | Approximately 2 Years
  The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Part 1 and 2: Volume of Distribution at Steady-State (Vss) of Duvortuxizumab | Approximately 2 Years
  The Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of duvortuxizumab at steady state.
Part 1 and 2: Immunogenicity of Duvortuxizumab | Approximately 2 Years
  Plasma levels of antibodies to duvortuxizumab for evaluation of potential immunogenicity.
Part 2: Duration of Response (DoR) | Approximately 2 Years
  The DoR is defined as the time from the first observed response (CR or PR) to documented disease progression or death due to any cause.
Part 2: Progression Free Survival (PFS) for DLBCL, FL, MCL, and CLL | Approximately 2 Years
  The PFS is defined as the time from date of the first dose of study drug to documented disease progression or death due to any cause.
Part 2: Percentage of Participants With Complete Response (CR) | Approximately 2 Years
  The CR is defined as a best response of CR according to the Criteria for Response Assessment of Non-Hodgkin Lymphomas (NHL), International Workshop on Chronic Lymphocytic Leukemia (CLL) or Response Criteria for acute lymphoblastic leukemia (ALL).
Part 2: Percentage of Participants with Overall Survival | Up to followup (Approximately 2 Years)
  Overall survival is defined as the duration from the date of the first dose of the study drug to the date of death for DLBCL, FL, MCL, CLL, and ALL.
Part 1 and 2: Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (Approximately 2 Years)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 2: Relapse-Free survival for Acute Lymphoblastic Leukemia (RFS for ALL) | Approximately 2 Years
  Relapse free survival (RFS) is defined as time from the date of the first dose of the study drug to relapse from CR, progressive disease, or death due to any cause for ALL.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (6):
  - Detroit, Michigan
  - New York, New York
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
- Belgium (3):
  - Edegem
  - Leuven
  - Wilrijk
- France (4):
  - Lille
  - Pierre-Bénite
  - Rennes
  - Tours
- Israel (4):
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Spain (3):
  - Barcelona
  - Madrid
  - Salamanca